CLINICAL TRIAL: NCT02291016
Title: A Randomized, Double-Dummy, Crossover, Single-Center Study Comparing the Efficacy of Nebulizers Versus Dry Powder Inhalers in the Treatment of Patients Recovering From Severe Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: COPD Aerosol Study Comparing the Efficacy of Nebulizers Versus Dry Powder Inhalers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Collaborators: Mylan Specialty L.P. (Unknown)
Responsible Party: Principal Investigator, Rajiv Dhand, MD, Principal Investigator, University of Tennessee Graduate School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 3798
Record Dates: First submitted 2014-11-05; First posted 2014-11-14 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: COPD Exacerbation
Keywords: COPD; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formoterol via DPI then Formoterol via nebulizer (Active Comparator): Group A: Received Formoterol 12 µg via DPI and placebo via nebulizer at treatment visit #1, and Formoterol 20 µg (solution form) via nebulizer and placebo via DPI at treatment visit 2.
  Placebo: The placebo used will be sterile, preservative free, normal saline for nebulizer inhalation and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
  Interventions: Drug: Formoterol; Other: Placebo
- Formoterol via nebulizer then Formoterol via DPI (Active Comparator): Group B: Received Formoterol 20 µg (solution form) via nebulizer and placebo via a DPI at treatment visit #1, and Formoterol 12 µg via a DPI with placebo via nebulizer at treatment visit 2.
  Placebo: The placebo used will be sterile, preservative free, normal saline for nebulizer inhalation and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
  Interventions: Drug: Formoterol; Other: Placebo

INTERVENTIONS:
Drug: Formoterol — Comparison of dosage administered via a nebulizer versus dosage administered via a dry powder inhaler. 12 µg Formoterol with the dry powder inhaler and 20 µg (solution form) of Formoterol with the nebulizer. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
  Other Names: Foradil; PERFOROMIST
Other: Placebo — Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
  Other Names: Normal Saline

SUMMARY:
The purpose of this study is to compare drug delivery and lung function after treatment with formoterol from a nebulizer versus a dry powder inhaler (DPI) in patients recovering from severe exacerbations of COPD. This is to determine if one device is superior in providing better lung function and drug deposition in this clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Current or past cigarette smoking history of >/= 10 pack-years.
* FEV1/FVC ratio </= 70%.
* Known diagnosis of COPD.
* Current hospitalization for a primary diagnosis of acute exacerbation of COPD.
* Must be able to understand and willing to sign an informed consent document.

Exclusion Criteria:

* On a ventilator or mask ventilation.
* Allergy or contraindication to Formoterol use.
* Marked QTc prolongation (> 450 ms).
* Liver cirrhosis or chronic renal insufficiency (serum creatinine > 2 mg/dL).
* Atrial fibrillation with rapid ventricular response (heart rate > 110 bpm) or ventricular arrhythmia (frequent PVCs, ventricular tachycardia).
* Acute myocardial infarction within 12 weeks of patient study registration.
* Known pulmonary embolism.
* Known or suspected lung cancer.
* Known neuromuscular disease, stroke with residual hemiparesis, or untreated Parkinsonism
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices, diaphragm, or sub dermal implants).
* Inability to understand instructions.
* Participation in another investigational drug clinical trial within 30 days of patient study registration.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Dhand, MD, Principal Investigator — University of Tennessee Medical Center
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Formoterol Via DPI Then Formoterol Via Nebulizer: Group A: Received Formoterol 12 µg via DPI and placebo via nebulizer at treatment visit #1, and then Formoterol 20 µg (solution form) via nebulizer and placebo via DPI at treatment visit 2.
  Placebo: Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
- Formoterol Via Nebulizer Then Formoterol Via DPI: Group B: Received Formoterol 20 µg (solution form) via nebulizer and placebo via a DPI at treatment visit #1, and then Formoterol 12 µg via a DPI with placebo via nebulizer at treatment visit 2.
  Placebo: Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
Period: Visit 1
Arm/Group | Formoterol Via DPI Then Formoterol Via Nebulizer | Formoterol Via Nebulizer Then Formoterol Via DPI
Started | 2 | 5
Completed | 2 | 5
Not Completed | 0 | 0
Period: Visit 2
Arm/Group | Formoterol Via DPI Then Formoterol Via Nebulizer | Formoterol Via Nebulizer Then Formoterol Via DPI
Started | 2 | 5
Completed | 1 (Patients did not meet visit 2 FEV1 criteria ( 15% or closer to value at visit 1)) | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Seven total subjects were studied. Order of crossover dosing as follows:
  Randomization:
  Group A:formoterol via DPI/placebo via nebulizer visit 1, and formoterol via nebulizer/placebo via DPI at visit 2.
  Group B:formoterol via nebulizer/placebo via a DPI at visit 1, and formoterol via DPI/placebo via nebulizer at visit 2.
Groups:
- Formoterol Via DPI Then Formoterol Via Nebulizer: Group A: Received Formoterol 12 µg via DPI and placebo via nebulizer at treatment visit #1, and Formoterol 20 µg (solution form) via nebulizer and placebo via DPI at treatment visit 2.
  Placebo: Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
- Formoterol Via Nebulizer Then Formoterol Via DPI: Group B: Received Formoterol 20 µg (solution form) via nebulizer and placebo via a DPI at treatment visit #1, and Formoterol 12 µg via a DPI with placebo via nebulizer at treatment visit 2.
  Placebo: Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
- Total: Total of all reporting groups
Arm/Group | Formoterol Via DPI Then Formoterol Via Nebulizer | Formoterol Via Nebulizer Then Formoterol Via DPI | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (3.6) | 61.2 (8.3) | 61.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between the Values of Area Under the Response Curve for FEV1
Description: The difference between the values of area under the response curve for FEV1 from baseline through four hours (AUC FEV1 0-4h) after inhalation of formoterol with a nebulizer or a dry powder inhaler.
Time Frame: Baseline through study completion (visit 1 through visit 2)
Population: Participants who received a dose of formoterol via nebulizer AND formoterol via dry powder were included. One patient did not complete the full study, which is why only 6 participants who took formoterol with Nebulizer were analyzed. Collected at baseline, visit 1, and visit 2 at pre-dose then 30 minutes,1hr, 2hr, and 4hr post-dose
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Groups:
- Formoterol With Nebilizer and Placebo With DPI: One dose of Formoterol 20 µg (solution form) via nebulizer at either visit 1 or visit 2 depending on group randomization, which is listed below.
  Randomization:
  Group A: Received formoterol via DPI and placebo via nebulizer at treatment visit #1, and formoterol via nebulizer and placebo via DPI at treatment visit 2.
  Group B: Received formoterol via nebulizer and placebo via a DPI at treatment visit #1, and formoterol via a DPI with placebo via nebulizer at treatment visit 2.
  Placebo: Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
- Formoterol With Dry Powder Inhaler: Formoterol: One dosing of 12 µg via dry powder inhaler at either visit 1 or visit 2 depending on randomization assignment, which is detailed below.
  Randomization:
  Group A: Received formoterol via DPI and placebo via nebulizer at treatment visit #1, and formoterol via nebulizer and placebo via DPI at treatment visit 2.
  Group B: Received formoterol via nebulizer and placebo via a DPI at treatment visit #1, and formoterol via a DPI with placebo via nebulizer at treatment visit 2.
  Placebo: Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
Arm/Group | Formoterol With Nebilizer and Placebo With DPI | Formoterol With Dry Powder Inhaler
Number analyzed (Participants) | 6 | 7
mcg*hr/mL | 203.0 (77.2) | 185.0 (84.0)

2. Secondary Outcome: Percentage Change in Peak FEV1 From Baseline After Inhalation of Formoterol
Description: Change in peak FEV1 from Baseline. This will be completed at visit 1 and visit 2.
  Steps:
  1. A baseline (pre-dose formoterol) FEV1 will be recorded.
  2. Subjects will be dosed with formoterol.
  3. Serial FEV1 assessments will completed at 15 minutes, 30 minutes, 1 hour, 2 hour, and 4 hour post dose of formoterol so a peak measurement can be recorded.
  4. A percentage of change between the baseline and peak FEV1 will be recorded for this outcome measure. A higher value indicates a better result.
Time Frame: From pre-dose formoterol (baseline 0hrs) to 30 minutes, 1,2, and 4 hours post dose at visit 1 and measured again at visit 2
Population: Participants who received a dose of formoterol via nebulizer AND formoterol via dry powder were included. One patient did not complete the full study, which is why only 6 participants who took formoterol with Nebulizer were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Formoterol With Dry Powder Inhaler and Placebo With Nebulizer: Formoterol: One dosing of 12 µg via dry powder inhaler at either visit 1 or visit 2 depending on randomization assignment, which is detailed below.
  Randomization:
  Group A: Received formoterol via DPI and placebo via nebulizer at treatment visit #1, and formoterol via nebulizer and placebo via DPI at treatment visit 2.
  Group B: Received formoterol via nebulizer and placebo via a DPI at treatment visit #1, and formoterol via a DPI with placebo via nebulizer at treatment visit 2.
  Placebo: Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
Arm/Group | Formoterol With Nebilizer and Placebo With DPI | Formoterol With Dry Powder Inhaler and Placebo With Nebulizer
Number analyzed (Participants) | 6 | 7
percent change | 28.2 (12.3) | 21.1 (23.4)

3. Secondary Outcome: Absolute Increase in FEV1 From Baseline After Inhalation of Formoterol
Description: Increase in FEV1 from Baseline to 4 hours post dose of formoterol. This will be completed at visit 1 and visit 2.
  Steps:
  1. A baseline (pre-dose formoterol) FEV1 was recorded.
  2. Subjects was dosed with formoterol.
  3. Serial FEV1 assessments were completed, and recorded at 15 minutes, 30 minutes, 1 hour, 2 hour, and 4 hour post dose of formoterol so serial FEV1 measurements could be recorded.
Time Frame: Measured at visit 1 and visit 2 after dosing and all FEV1 testing has been completed
Population: Participants who received a dose of formoterol via nebulizer AND formoterol via dry powder were included.One patient did not complete the full study, which is why only 6 participants who took formoterol with Nebulizer were analyzed.
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | Formoterol With Nebilizer and Placebo With DPI | Formoterol With Dry Powder Inhaler and Placebo With Nebulizer
Number analyzed (Participants) | 6 | 7
L/sec | 12.2 (7.1) | 9.5 (10.4)

4. Secondary Outcome: Peak FEV1 Between the Two Devices (Nebulizer and DPI)
Description: Change in peak FEV1 from Baseline. This will be completed at visit 1 and visit 2.
  Steps:
  1. A baseline (pre-dose formoterol) FEV1 was recorded.
  2. Subjects were dosed with formoterol.
  3. Serial FEV1 assessments were completed at 15 minutes, 30 minutes, 1 hour, 2 hour, and 4 hour post dose of formoterol so a peak measurement could recorded.
  5. Peak measurements from visit 1 and visit 2 will be compared for any significant change in FEV1 values.
Time Frame: Measured from Start of visit 1 until the completion of visit 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | Formoterol With Nebilizer and Placebo With DPI | Formoterol With Dry Powder Inhaler and Placebo With Nebulizer
Number analyzed (Participants) | 6 | 7
L/sec | 12.2 (7.1) | 9.5 (10.4)

5. Secondary Outcome: Change in FEV1 as a Percentage of Predicted Normal After Inhalation of Formoterol
Description: Change in FEV1 from Baseline through 4 hours post formoterol dose. This was completed at visit 1 and visit 2.
  Steps:
  1. A baseline (pre-dose formoterol) FEV1 was recorded.
  2. Subjects were dosed with formoterol.
  3. Serial FEV1 assessments were completed at 15 minutes, 30 minutes, 1 hour, 2 hour, and 4 hour post dose of formoterol and serial FEV1 values were recorded.
  4. A percentage of change from baseline FEV1 to each serial measurement of FEV1 was collected. The % of change at each time point was then used to get a measure of overall percentage change of the predicted FEV1 value.
Time Frame: Baseline through study completion (visit 1 through visit 2)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change of % predicted FEV1
Arm/Group | Formoterol With Nebilizer and Placebo With DPI | Formoterol With Dry Powder Inhaler and Placebo With Nebulizer
Number analyzed (Participants) | 6 | 7
percentage change of % predicted FEV1 | 21.5 (11.8) | 18.4 (14.9)

6. Secondary Outcome: Area Under the Response Curve for FVC From Baseline Through Four Hours (AUC FVC0-4h) After Inhalation of Formoterol
Description: Steps:
  1. A baseline (pre-dose formoterol) FVC was recorded.
  2. Subjects were dosed with formoterol.
  3. Serial FVC assessments were completed at 15 minutes, 30 minutes, 1 hour, 2 hour, and 4 hour post dose of formoterol and serial FVC values were recorded.
  Data was all time points were used to obtain the total area under the curve
Time Frame: Measured at visit 1 and again at the end of visit 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Formoterol With Nebilizer and Placebo With DPI | Formoterol With Dry Powder Inhaler and Placebo With Nebulizer
Number analyzed (Participants) | 6 | 7
mcg*hr/mL | 327.0 (75.0) | 293.4 (49.8)

7. Secondary Outcome: Percentage Change in Peak FVC From Baseline After Inhalation of Formoterol
Description: 1. A baseline (pre-dose formoterol) FVC was recorded.
  2. Subjects were dosed with formoterol.
  3. Serial FVC assessments were completed at 15 minutes, 30 minutes, 1 hour, 2 hour, and 4 hour post dose of formoterol and serial FVC values were recorded.
  4. A percentage of change between the baseline and peak FVC will be recorded for this outcome measure.
Time Frame: Measured at visit 1 and again at the end of visit 2
Population: Participants who received a dose of formoterol via nebulizer AND formoterol via dry powder were included.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Formoterol With Nebilizer and Placebo With DPI | Formoterol With Dry Powder Inhaler and Placebo With Nebulizer
Number analyzed (Participants) | 6 | 7
percent change | 22.1 (11.7) | 18.2 (13.0)

8. Secondary Outcome: Peak FVC Between the Two Devices (Nebulizer and DPI)
Description: Steps:
  1. A baseline (pre-dose formoterol) FVC was recorded.
  2. Subjects were dosed with formoterol.
  3. Serial FVC assessments were completed at 15 minutes, 30 minutes, 1 hour, 2 hour, and 4 hour post dose of formoterol and serial FVC values were recorded.
  4. Peak FVC was recorded for this outcome measure and compared amongst groups.
Time Frame: Peak FVC at visit 1 will be compared to the peak FVC at visit 2 for any significant change.
Population: Participants who received a dose of formoterol via nebulizer AND formoterol via dry powder were included.
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | Formoterol With Nebilizer and Placebo With DPI | Formoterol With Dry Powder Inhaler and Placebo With Nebulizer
Number analyzed (Participants) | 6 | 7
L/sec | 86.7 (22.0) | 82.0 (12.6)

9. Secondary Outcome: Change in Dyspnea Based on the Borg Dyspnea Scale for Shortness of Breath (Pre-dose Administration and 60 Minutes After Inhalation of Formoterol With a Nebulizer or a DPI)
Description: The Shortness of Breath Modified Borg Dyspnea Scale The scale goes from 0-10, zero meaning no difficulty breathing and ten meaning maximal difficulty. A decrease of score indicates an improvement. Patients were asked to complete the scale pre-dose and again one hour post formoterol dose. This was completed at both visit 1 and visit 2. The value recorded was the difference between the baseline value and the post 60 minute value.
Time Frame: Measured at visit 1 and again at the end of visit 2
Population: Participants who received a dose of formoterol via nebulizer AND formoterol via dry powder were included.
Measure: Mean (Standard Deviation); unit: change in score
Arm/Group | Formoterol With Nebilizer and Placebo With DPI | Formoterol With Dry Powder Inhaler and Placebo With Nebulizer
Number analyzed (Participants) | 6 | 7
change in score | -0.59 (0.63) | 0 (.50)

ADVERSE EVENTS:
Time Frame: Collected from subject randomization through subject study completion (visit 1-visit 2), which was approximately 9 days total.
Description: Instead of reporting the findings from Group A ( Dosed with Nebulizer placebo and DPI formoterol at visit 1, and dosed with nebulizer formoterol and DPI placebo at visit 2), and Group B (Dosed with nebulizer formoterol and DPI placebo at visit 1 , and dosed with nebulizer placebo and DPI formoterol at visit 2), we reported the adverse event groups by the following: Formoterol via Nebulizer and Formoterol via DPI, as patients were given both in this cross-over study.
Groups:
- Formoterol With Nebulizer: One dose of Formoterol 20 µg (solution form) via nebulizer at either visit 1 or visit 2 depending on group randomization, which is listed below.
  Randomization:
  Group A: Received formoterol via DPI and placebo via nebulizer at treatment visit #1, and formoterol via nebulizer and placebo via DPI at treatment visit 2.
  Group B: Received formoterol via nebulizer and placebo via a DPI at treatment visit #1, and formoterol via a DPI with placebo via nebulizer at treatment visit 2.
  Placebo: Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
- Formoterol With Dry Powder Inhaler: One dose of Formoterol 12 µg (solution form) via DPI at either visit 1 or visit 2 depending on group randomization, which is listed below.
  Randomization:
  Group A: Received formoterol via DPI and placebo via nebulizer at treatment visit #1, and formoterol via nebulizer and placebo via DPI at treatment visit 2.
  Group B: Received formoterol via nebulizer and placebo via a DPI at treatment visit #1, and formoterol via a DPI with placebo via nebulizer at treatment visit 2.
  Placebo: Comparison of drug administered via a nebulizer versus a dry powder inhaler. The placebo used will be sterile, preservative free, normal saline for inhalation for the nebulizer and a matched capsule without active drug for the dry powder inhaler. All patients will receive 2 ml of normal saline with the nebulizer to match the volume of nebulized formoterol solution. Patients will receive formoterol and placebo at both study visit #1 and visit #2.
Arm/Group | Formoterol With Nebulizer | Formoterol With Dry Powder Inhaler
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No